CLINICAL TRIAL: NCT02743325
Title: Optimisation of Catheter Navigation With As Low As Reasonable Achievable Fluoroscopy for Amelioration of Ablation Success in Patients With SupraVentricular Tachycardia (ALARA-SVT)
Brief Title: As Low As Reasonable Achievable Fluoroscopy for SVT Ablation
Acronym: ALARA-SVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Kobza (Other)
Responsible Party: Sponsor-Investigator, Richard Kobza, PD Dr. med., Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-142
Record Dates: First submitted 2016-03-15; First posted 2016-04-19 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Symptomatic Supraventricular Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALARA protocol (Active Comparator): SVT ablation by ALARA protocol
  Interventions: Procedure: SVT ablation by ALARA protocol
- current treatment (Active Comparator): SVT ablation by conventional protocol
  Interventions: Procedure: SVT ablation by conventional protocol

INTERVENTIONS:
Procedure: SVT ablation by ALARA protocol — Catheter ablation is a procedure that uses radiofrequency energy (similar to microwave heat) to destroy a small area of heart tissue that is causing arrhythmias. Destroying this tissue helps restore your heart's regular rhythm. The usage of CartoUnivuTM allows a seamless combination of a fluoro image and Carto® 3 System maps into a single view.
  Other Names: radiofrequency ablation by ALARA protocol
  Arms: ALARA protocol
Procedure: SVT ablation by conventional protocol — Catheter ablation is a procedure that uses radiofrequency energy (similar to microwave heat) to destroy a small area of heart tissue that is causing arrhythmias. Destroying this tissue helps restore your heart's regular rhythm. The convention Ablation procedure works without a 3D navigation System.
  Other Names: radiofrequency ablation by conventional protocol
  Arms: current treatment

SUMMARY:
Supraventricular tachycardia ablations of the Conformité Européenne (CE)-certified (since 2013) CartoUnivuTM module (Biosense Webster, Diamond Bar, USA) allows a seamless combination of a fluoro image and Carto® 3 System maps into a single view. This helps to reduce fluoroscopy levels and reduce exposure time for physicians, staff and patients to as low as reasonably achievable. The UnivuTM technology will be compared in a randomized manner to the conventional radiofrequency Ablation.

DETAILED DESCRIPTION:
Aim of the current Randomized Clinical Study is to assess the safety and efficiency in supraventricular tachycardia ablations of the CE-certified (since 2013) CartoUnivuTM module (Biosense Webster, Diamond Bar, USA), allowing a seamless combination of a fluoro Image and Carto® 3 System maps into a single view. It helps reduce fluoroscopy levels - consistent with the ALARA principle of reducing exposure for physicians, staff and patients to as low as reasonably achievable. The UnivuTM technology will be compared in a randomized manner to the conventional radiofrequency (RF) ablation.

Patients with symptomatic supraventricular tachycardia (SVT) will be included, more specifically patients with atrioventricular nodal re-entrant tachycardia (AVRNT), atrioventricular re-entrant tachycardia (AVRT) and typical atrial flutter (TAF). Current ablative treatment consists in destroying small areas of myocardial tissue or conduction system, or both, that are critical to the initiation or maintenance of the arrhythmia (slow pathway Ablation in the case of AVRNT, anomalous extra nodal connections between the atrium and ventricle along the atrioventricular groove in AVRT and cavo-tricuspid isthmus in the case of TAF).

However, SVT ablations without a 3D navigation system have a certain fluoroscopy time and radiation exposure, respectively. Prolonged fluoroscopy and radiation exposure during ablation may potentially cause an increase in the lifetime risk of fatal malignancy.

In a 1-year follow-up the arrhythmia recurrence rate without anti-arrhythmic drugs will be assessed using 7-day holter recording in 60 patients undergoing CartoUnivuTM guided SVT ablation (group A) vs. 60 patients undergoing conventional RF-catheter ablation (without CartoUnivuTM, group B).

All patients will stop anti-arrhythmic drugs at least 1 week before the date of ablation. Each patient will undergo transthoracal echocardiography (TTE) before the intervention. In case transseptal is needed, heparin will be administered after successful transseptal puncture with an activated clotting time (ACT)-target ≥325 sec.

Following data will be acquired:

* Age, gender, presence of structural heart disease (SHD), co-morbidities
* Duration of arrhythmia (first manifestation and longest lasting episode)
* Current and failed antiarrhythmic therapy
* Echocardiography: Dilatation, hypertrophy, regurgitation, Left ventricular ejection fracture (LVEF), any important other abnormalities (e.g. prolapse)

Ablation for SVT:

The following concept will be used for ablation of the slow pathway ablation in the case of AVRNT, anomalous extra nodal connections between the atrium and ventricle along the atrioventricular groove in AVRT and cavo-tricuspid isthmus in the case of TAF: Using the 3D-electro-anatomic system (CARTO3®) with the module for fluoroscopy integration (UnivuTM), the diagnostic catheters (10 poles deflectable catheter and fixed 4 poles catheter) will be introduced without using fluoroscopy after the registration phase and the transfer of a fluoroscopic image in anteroposterior (AP) and left anterior oblique (LAO) projections into the Carto3® System.

Once the electrophysiology study is realized and the arrhythmia identified (an activation can be used for this purpose), the ablation catheter (Navistar® 4mm/8mm, Biosense Webster, Diamond Bar, USA) is then introduced (also without the use of fluoroscopy). In case no map was done for local activation time information, specific tags will be taken:

* AVRNT: His, coronary Sinus (CS) ostium
* AVRT
* right atrium: His, CS ostium, tricuspid annulus
* left atrium: left inferior vein, appendage, mitral annulus
* AF: His, ostium of the inferior vena cava, tricuspid annulus

Aim of the ablation procedure is to ablate small areas of myocardial tissue or conduction system, or both, that are critical to the initiation or maintenance of the arrhythmia (slow pathway ablation in the case of AVRNT, anomalous extra nodal connections between the atrium and ventricle along the atrioventricular groove in AVRT and cavo-tricuspid isthmus in the case of TAF) using the CartoUnivuTM module (Biosense Webster, Diamond Bar, USA) for fluoroscopy integration on the Carto 3® System, with no further arrhythmia inducibility.

If a non-clinical arrhythmia corresponding to the patient symptoms is induced, pharmacological and/or electrical cardioversion in to sinus rhythm will be performed. If a coronariography is performed, the procedure time, fluoroscopy time and doses used will be discounted from the overall respective measurements.

Annotation of ablation sites on the 3D-map must be performed only by the VisiTag algorithm (integrated in the CARTO3® system), which will allow post-procedural analysis of catheter stability at each RF delivery site, duration of RF-application values and catheter stability during ablation.

The following procedural data will be acquired:

* Total procedure time (femoral vein puncture until removement of sheaths)
* Use of long sheath for ablation catheter (name and type, steerable or not)
* Duration of RF-delivery and mean delivered RF-power
* Fluoroscopy duration and doses
* Activation map: yes/no, how many points
* Complications

Follow-up:

* Number of patients with arrhythmia recurrence after blanking period (3months post 1st ablation procedure and stop of antiarrhythmic drugs)
* 7-day holter for rhythm monitoring at 6 and 12 months
* Phone contact / questionnaire to document patients symptoms and medications after 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic SVT undergoing first SVT ablation procedure (and no prior history of cardiac surgery
* Structurally normal heart (no major cardiac defects)

Exclusion Criteria:

* Previous ablation for SVT (or cardiac surgery)
* Contra-indications to catheter ablation therapy
* Congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
recurrence of arrhythmia documented by ECGs | within 90 days after the ablation procedure
  Documentation by ECG,7-day-holter ECG, symptoms description by the patient

SECONDARY OUTCOMES:
total fluoroscopy time in minutes | during the ablation procedure
  fluoroscopy time measured in minutes administered during the Ablation procedure
total radiation exposure in gy | during the ablation procedure
  Exposition of the Patient to Radiation during the ablation procedure measured in gy
Duration of Ablation procedure in minutes | skin to skin of the ablation procedure
  time needed to complete the procedure
Composite adverse events | within the first 30 days post ablation procedure
  Death of any cause, bleeding, vascular complications, and high-degree atrioventricular block

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kobza, PD Dr. med., Principal Investigator — Luzerner Kantonsspital

IPD SHARING:
Plan to Share IPD: No